CLINICAL TRIAL: NCT01606423
Title: The Effect of LY2409021 on Blood Glucose Concentrations During Hyperglucagonaemia in Healthy Male Subjects
Brief Title: The Effect of LY2409021 on Blood Sugar Levels When Glucagon Levels Are Increased in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 11165; I1R-FW-GLBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — adomeglivant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Administered once, orally
  Interventions: Drug: Placebo
- 10 mg LY2409021 (Experimental): 10 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- 22.5 mg LY2409021 (Experimental): 22.5 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- 60 mg LY2409021 (Experimental): 60 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- 200 mg LY2409021 (Experimental): 200 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- 500 mg LY2409021 (Experimental): 500 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: Placebo — Administered orally, single dose
  Arms: Placebo
Drug: LY2409021 — Administered orally, single dose
  Arms: 10 mg LY2409021; 200 mg LY2409021; 22.5 mg LY2409021; 500 mg LY2409021; 60 mg LY2409021

SUMMARY:
This is a study to measure the effect that various doses of LY2409021 have on blood sugar levels and on the amount of glucose released by the liver, when glucagon is given to increase these. Each participant may receive up to 2 single doses of LY2409021 in 2 different study periods, with a minimum 13-day washout between dosing periods. This study is approximately 9 weeks long, not including screening. A screening appointment is required within 6 weeks prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be a healthy male
* Have a screening body mass index (BMI) of 18.5 to 29.9 kg/m^2 inclusive
* Have a fasting blood glucose between 3.0-6.0 millimoles/liter (mmol/L) (inclusive) at screening

Exclusion Criteria:

* Are allergic to LY2409021, insulin, glucagon, somatostatin, or similar drugs
* Have a regular alcohol intake greater than 21 units/week, or are unwilling to stop alcohol as required by the study restrictions (1 unit = 360 mL of beer, or 150 mL of wine, or 45 mL of spirits)
* Are currently smokers or have used tobacco products on a regular basis in the 6 months prior to screening
* Have received any medication known to affect glucose metabolism in the 1 month before the study
* Have a significant blood disorder and/or donated blood (450 mL or more) in the last 3 months

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Maximum glucose response during a 3-hour glucagon infusion | During a 3-hour glucagon infusion

SECONDARY OUTCOMES:
Total glucose released from the liver during a 3-hour glucagon infusion | During a 3-hour glucagon infusion
Maximum glucose release from the liver during a 3-hour glucagon infusion | During a 3-hour glucagon infusion

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore